CLINICAL TRIAL: NCT03724396
Title: Novel Executive Function Training for Obesity
Acronym: NEXT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Dawn Eichen, Assistant Adjunct Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K23DK114480 (NIH); K23DK114480 (NIH)
Record Dates: First submitted 2018-10-25; First posted 2018-10-30 (Actual); Results first posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Overweight and Obesity
Keywords: weight loss; executive function
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novel Executive Function Training - NEXT (Experimental): Same as BWL with some additional strategies targeted at improving executive function to help adherence to BWL skills.
  Interventions: Behavioral: Behavioral Weight Loss - BWL; Behavioral: Novel Executive Function Training - NEXT
- Behavioral Weight Loss - BWL (Active Comparator): All participants will be instructed on how to consume a balanced deficit diet of conventional foods; individual goals for energy intake will be based on initial body weight. Participants will be instructed in measuring portion sizes, counting calories (with a calorie counter provided or on their phone), and self-monitoring food intake. The physical activity program will focus on increasing both lifestyle activity and structured exercise programs. Behavior change recommendations include stimulus control, self-monitoring, goal setting, managing high-risk situations, meal planning, slowing eating, problem solving, social support, cognitive restructuring, lapse and relapse prevention skills, and maintaining weight loss.
  Interventions: Behavioral: Behavioral Weight Loss - BWL

INTERVENTIONS:
Behavioral: Behavioral Weight Loss - BWL — All participants will be instructed on how to consume a balanced deficit diet of conventional foods; individual goals for energy intake will be based on initial body weight. Participants will be instructed in measuring portion sizes, counting calories (with a calorie counter provided or on their phone), and self-monitoring food intake. The physical activity program will focus on increasing both lifestyle activity and structured exercise programs. Behavior change recommendations include stimulus control, self-monitoring, goal setting, managing high-risk situations, meal planning, slowing eating, problem solving, social support, cognitive restructuring, lapse and relapse prevention skills, and maintaining weight loss.
Behavioral: Novel Executive Function Training - NEXT — Modifies programs like CogSMART and cognitive remediation training to help participants improve executive functioning to adhere to recommendations from BWL.
  Arms: Novel Executive Function Training - NEXT

SUMMARY:
Currently, the best behavioral treatments for obesity only work for 50% of adults, and of those who initially succeed, most do not maintain their weight loss. One reason for this failure may be due to neurocognitive deficits found among individuals with obesity, particularly related to executive function, which make it difficult for these adults to adhere to treatment recommendations. The proposed study aims to develop a Novel Executive Function Treatment (NEXT), which when administered prior to the behavioral treatment, could help improve outcomes by addressing the neurocognitive deficits in adults with overweight or obesity.

DETAILED DESCRIPTION:
First, to assist with treatment development, two groups of approximately 10 participants will be enrolled in a 12-week open-label treatment group of NEXT. These participants will then provide qualitative feedback to help with treatment development. After the two pilot groups, a randomized control trial will evaluate NEXT compared to standard BWL to assess feasibility, acceptability and preliminary efficacy. Treatment will be 6 months long and assessments will occur at baseline, mid-treatment, post-treatment and 6-months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Ability to read English at a 6th grade level
* BMI >25 and ≤45
* Difficulties with executive functioning

Exclusion Criteria:

* Medical condition that requires physician monitoring to participate in weight control program or prohibits safely participating in recommended physical activity
* Psychiatric condition that could interfere with program participant (e.g., substance abuse, suicide attempt within previous 6 months, active purging)
* Currently pregnant, lactating or plan to be in the timespan of program follow-up
* Current enrollment in an organized weight control program
* Change in psychotropic medication or other medication that could have impact on weight during the previous 3 months
* History of bariatric surgery
* History of learning disorder, neurological condition or injury

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2023-01-14 (Actual); Study Completion 2023-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Eichen, PhD, Principal Investigator — UC San Diego
Locations (1):
- UCSD Center for Healthy Eating and Activity Research (CHEAR, La Jolla, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Novel Executive Function Training - NEXT | Behavioral Weight Loss - BWL
Started | 34 | 33
Mid Treatment | 33 | 32
Post-Treatment | 32 | 31
6-month Follow-up | 32 | 32
Completed | 32 | 32
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Novel Executive Function Training - NEXT | Behavioral Weight Loss - BWL | Total
Number analyzed (Participants) | 34 | 33 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (11.0) | 44.6 (13.3) | 45.8 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 27 | 56
  Male | 5 | 6 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 13
  Not Hispanic or Latino | 27 | 27 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 6 | 5 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 22 | 20 | 42
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Feasibility as Measured by Attendance
Description: Number of Treatment Sessions Attended
Time Frame: Over the course of 6 months of treatment
Population: total intention to treat sample evaluated
Measure: Median (Inter-Quartile Range); unit: Sessions
Arm/Group | Novel Executive Function Training - NEXT | Behavioral Weight Loss - BWL
Number analyzed (Participants) | 34 | 33
Sessions | 18 [17 to 19] | 18 [16 to 19]

2. Primary Outcome: Acceptability
Description: Ratings of usefulness of treatment
Time Frame: At 6 months
Population: Includes all participants who responded to the acceptability survey at post-treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Novel Executive Function Training - NEXT | Behavioral Weight Loss - BWL
Number analyzed (Participants) | 31 | 30
Participants
  Strongly Agreed or Agreed that treatment helped develop healthy habits | 25 | 26
  Strongly Agreed or Agreed that they would recommend the program to a friend | 28 | 24

3. Other Pre Specified Outcome: BMI Change
Description: change in BMI (kg/m2)
Time Frame: From baseline through mid-treatment (3 months), post-treatment (6 months), and 6-month follow-up (12 months)
Population: All available data were used but at some timepoints data was missing. Numbers analyzed represent number of individuals providing data at each timepoint.
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Novel Executive Function Training - NEXT | Behavioral Weight Loss - BWL
Number analyzed (Participants) | 34 | 33
kg/m2
  Baseline BMI | 33.3 (4.3) | 33.2 (5.5)
  Mid-Treatment BMI: number analyzed (Participants) | 33 | 32
  Mid-Treatment BMI | 32.6 (4.4) | 32.5 (5.6)
  Post-Treatment BMI: number analyzed (Participants) | 32 | 31
  Post-Treatment BMI | 32.0 (4.8) | 31.7 (5.8)
  6-Month Follow-up BMI: number analyzed (Participants) | 32 | 32
  6-Month Follow-up BMI | 32.4 (4.7) | 33.1 (6.5)

4. Other Pre Specified Outcome: Executive Function
Description: Change in executive function measured by Behavior Rating Inventory of Executive Function- Adult Version (BRIEF-A) Global Executive Composite T score which reflects overall levels of executive dysfunction; T-scores have a mean of 50 and a standard deviation of 10. Higher T-scores mean greater executive dysfunction or lower/poorer executive function. T-scores at or greater than 65 are considered clinically significant measure of executive dysfunction.
Time Frame: From baseline through mid-treatment (3 months), post-treatment (6 months), and 6-month follow-up (12 months)
Population: Numbers per row represent numbers of individual providing data for this specific measure at each timepoint. All analyses conducted are intent to treat framework.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Novel Executive Function Training - NEXT | Behavioral Weight Loss - BWL
Number analyzed (Participants) | 34 | 33
T-score
  Baseline GEC | 57.4 (12.7) | 57.2 (12.5)
  Mid-Treatment GEC: number analyzed (Participants) | 33 | 32
  Mid-Treatment GEC | 58.1 (12.9) | 55.3 (11.2)
  Post-Treatment GEC: number analyzed (Participants) | 31 | 30
  Post-Treatment GEC | 56.1 (13.7) | 59.5 (11.7)
  6-Month Follow-up GEC: number analyzed (Participants) | 29 | 29
  6-Month Follow-up GEC | 57.1 (13.0) | 59.2 (11.0)

ADVERSE EVENTS:
Time Frame: From baseline assessment through 6 months follow-up (~12 months)
Description: At each assessment timepoint following baseline (mid-treatment, post-treatment, and 6-month follow-up) participants were asked about any changes to medications and any changes to their health conditions/diagnoses
Arm/Group | Novel Executive Function Training - NEXT | Behavioral Weight Loss - BWL
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/33
Other Adverse Events (participants affected / at risk) | 0/34 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/96/NCT03724396/Prot_SAP_000.pdf